CLINICAL TRIAL: NCT06015477
Title: Stent-Assisted Coiling Followed by Ticagrelor Monotherapy Instead of Dual Antiplatelet Therapy in Endovascular Treatment of Unruptured Intracranial Aneurysm (SAC-TIDE) ---a Pilot Study
Brief Title: Stent-Assisted Coiling Followed by Ticagrelor Monotherapy Instead of Dual Antiplatelet Therapy in Unruptured Intracranial Aneurysm
Acronym: SAC-TIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAC-TIDE
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Intracranial Aneurysm; Stent Complication
Keywords: Intracranial Aneurysm; Stent-Assisted Coiling; Ticagrelor; Dual Antiplatelet
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: Patients meeting the enrollment criteria will be randomly assigned to one of the two treatment groups (1:1) and will be followed up for 1 year. All patients received oral clopidogrel 75 mg + aspirin 100 mg for 3-5 days preoperatively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ticagrelor monotherapy group (Experimental): Ticagrelor monotherapy (starting dose of ticagrelor was a single loading dose of 180mg (90mg x 2 tablets) and thereafter 1 tablet (90mg) each time, twice daily.). After 1 month, continuation to ticagrelor monotherapy for 1 year.
  Interventions: Drug: Ticagrelor monotherapy
- Dual Antiplatelet Therapy group (Active Comparator): Clopidogrel 75mg + Aspirin 100mg 1 month, after 1 month, change to aspirin 100mg 1 year.
  Interventions: Drug: Dual Antiplatelet Therapy

INTERVENTIONS:
Drug: Ticagrelor monotherapy — starting dose of ticagrelor was a single loading dose of 180mg (90mg x 2 tablets) and thereafter 1 tablet (90mg) each time, twice daily.
  Arms: ticagrelor monotherapy group
Drug: Dual Antiplatelet Therapy — Clopidogrel 75mg + Aspirin 100mg 1 month, after 1 month, change to aspirin 100mg 1 year.
  Arms: Dual Antiplatelet Therapy group

SUMMARY:
The primary goal of the trial is to investigate whether the experimental arms (receiving the P2Y12 inhibitor Ticagrelor) compared with the control arm (taking dual antiplatelet therapy) could reduce bleeding complications in patients with intracranial aneurysms undergoing Stent-Assisted Coiling.

DETAILED DESCRIPTION:
Bleeding complications associated with the use of DAPT have been of great concern, with up to one-third of PCI patients treated with DAPT previously reported to suffer from nuisance bleeding. Once any of these bleeding complications occur, adherence to the DAPT regimen may become difficult. Antiplatelet agents are necessary for patients undergoing stent-assisted spring coil embolisation of intracranial aneurysms and are key to reducing thrombosis leading to ischaemic stroke events in post-procedural patients.

Currently neither long-term DAPT nor short-duration DAPT followed by aspirin monotherapy is fully satisfactory. Patients with aneurysms without underlying intracranial atherosclerotic disease have relatively lower ischaemic risk factors, and antiplatelet medication after stenting remains to be improved. Ticagrelor monotherapy was associated with a lower risk of major bleeding and no measurable increase in ischaemic events after a short course of 1- or 3-month DAPT. The study indicated no difference in stroke or death between mono- and dual-antiplatelet therapy after carotid artery placement, and P2Y12 inhibitor monotherapy may be an effective strategy to reduce severe bleeding complications while preserving ischemic benefits for patients. This study investigates the comparative efficacy and safety of stent-assisted coiling therapy for intracranial aneurysms after ticagrelor monotherapy as an alternative to dual antiplatelet therapy, to reduce the incidence of bleeding complications in patients, and thus to improve the antiplatelet strategy after stent-assisted coiling therapy for intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a definitive diagnosis of an unruptured intracranial aneurysm with imaging suggestive of an aneurysm <10 mm
2. Patients who successfully underwent stent-assisted spring coil treatment for intracranial aneurysms without acute ischaemic or bleeding stroke events in the perioperative period
3. Age 18-60 years old
4. Patients with no previous history of chronic diseases such as hypertension, diabetes mellitus, coronary heart disease, hyperlipidaemia and so on
5. Agreed to participate in this study and gave informed consent for the collection and preservation of case data and the follow-up process.

Exclusion Criteria:

1. Planned surgery or intervention during the experiment requiring study drug discontinuation; (2) Contraindications requiring oral anticoagulation or aspirin or clopidogrel; (3) History of severe central nervous system damage (e.g., as a result of tumour, aneurysm, intracranial or spinal cord surgery); (4) Severe liver disease, including hepatic failure, cirrhosis, portal hypertension (oesophageal varices), active hepatitis; (5 ) severe renal dysfunction (creatinine more than 1.5 times the upper limit of the normal range); (6) severe heart failure (NYHA class:III ~ IV); high risk for chronic arrhythmias (1st or 2nd degree atrioventricular block due to sinus node disease, bradycardic syncope without pacemaker); diagnosis or suspected diagnosis of acute coronary syndrome; bacterial endocarditis, pericarditis; (7) severe comorbidities or patients with active cancer with a life expectancy of less than 2 years; (8) participation in another clinical study using an experimental product within the past 30 days; currently receiving an experimental drug or device; and (9) pregnant, currently pregnant, or of childbearing potential without birth control or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Hemorrhage | Within one year after surgery
  The incidence of bleeding defined by Bleeding Academic Research Consortium
Composite endpoint of all-cause mortality, cerebrovascular accident or urgent target vessel revascularization. | Within one year after surgery
  Co-Primary Efficacy Endpoint (non-inferiority hypothesis)

SECONDARY OUTCOMES:
ischemic stroke | This will be assessed during the first year of follow-up.
  ischemic stroke or death during 1 year of follow-up in an intention-to treat analysis.
Stent thrombosis | Within one year after surgery
  Stent thrombosis
BARC 1-5 type bleeding | Within one year after surgery
  bleeding defined by Bleeding Academic Research Consortium

CONTACTS AND LOCATIONS:
Overall Officials: Hua Lu, Doctor, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Hua Lu, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available to other researchers under the approval of the ethical committee.
Supporting Information: Study Protocol, CSR
Time Frame: the data will be available when summary data are published.

REFERENCES:
- [Result] Ben-Dor I, Torguson R, Scheinowitz M, Li Y, Delhaye C, Wakabayashi K, Maluenda G, Syed AI, Collins SD, Gonzalez MA, Gaglia MA Jr, Xue Z, Kaneshige K, Satler LF, Suddath WO, Kent KM, Pichard AD, Waksman R. Incidence, correlates, and clinical impact of nuisance bleeding after antiplatelet therapy for patients with drug-eluting stents. Am Heart J. 2010 May;159(5):871-5. doi: 10.1016/j.ahj.2010.01.016. PMID 20435198
- [Result] Kim KS, Fraser JF, Grupke S, Cook AM. Management of antiplatelet therapy in patients undergoing neuroendovascular procedures. J Neurosurg. 2018 Oct;129(4):890-905. doi: 10.3171/2017.5.JNS162307. Epub 2017 Dec 1. PMID 29192856
- [Result] Nordeen JD, Patel AV, Darracott RM, Johns GS, Taussky P, Tawk RG, Miller DA, Freeman WD, Hanel RA. Clopidogrel Resistance by P2Y12 Platelet Function Testing in Patients Undergoing Neuroendovascular Procedures: Incidence of Ischemic and Hemorrhagic Complications. J Vasc Interv Neurol. 2013 Jun;6(1):26-34. PMID 23826440
- [Result] Gutierrez J, Turan TN, Hoh BL, Chimowitz MI. Intracranial atherosclerotic stenosis: risk factors, diagnosis, and treatment. Lancet Neurol. 2022 Apr;21(4):355-368. doi: 10.1016/S1474-4422(21)00376-8. Epub 2022 Feb 7. PMID 35143758
- [Result] Valgimigli M, Mehran R, Franzone A, da Costa BR, Baber U, Piccolo R, McFadden EP, Vranckx P, Angiolillo DJ, Leonardi S, Cao D, Dangas GD, Mehta SR, Serruys PW, Gibson CM, Steg GP, Sharma SK, Hamm C, Shlofmitz R, Liebetrau C, Briguori C, Janssens L, Huber K, Ferrario M, Kunadian V, Cohen DJ, Zurakowski A, Oldroyd KG, Yaling H, Dudek D, Sartori S, Kirkham B, Escaned J, Heg D, Windecker S, Pocock S, Juni P; SIDNEY Collaboration. Ticagrelor Monotherapy Versus Dual-Antiplatelet Therapy After PCI: An Individual Patient-Level Meta-Analysis. JACC Cardiovasc Interv. 2021 Feb 22;14(4):444-456. doi: 10.1016/j.jcin.2020.11.046. PMID 33602441
- [Result] Jin Y, Huang H, Shu X, Chen S, Lu L, Gao X, Wu Z. P2Y12 inhibitor monotherapy and dual antiplatelet therapy after percutaneous coronary intervention: An updated meta-analysis of randomized trials. Thromb Res. 2021 Feb;198:115-121. doi: 10.1016/j.thromres.2020.11.038. Epub 2020 Dec 7. PMID 33316640